CLINICAL TRIAL: NCT01637961
Title: A Phase II Evaluation of MLN8237 (NSC# 747888) in the Treatment of Recurrent or Persistent Leiomyosarcoma of the Uterus
Brief Title: Alisertib in Treating Patients With Recurrent or Persistent Leiomyosarcoma of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01982; NCI-2012-01982 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0231D; CDR0000736350; GOG-0231D (Other: NRG Oncology); GOG-0231D (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Results first posted 2015-07-17 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Uterine Corpus Sarcoma; Uterine Corpus Leiomyosarcoma
MeSH Terms: interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (alisertib) (Experimental): Patients receive alisertib PO BID on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Alisertib — Given PO
  Other Names: Aurora A Kinase Inhibitor MLN8237; MLN-8237; MLN8237
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well alisertib works in treating patients with leiomyosarcoma of the uterus that has come back or persistent. Alisertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the clinical activity of MLN8237 (alisertib) in patients with recurrent or persistent leiomyosarcoma of the uterus who have received one or two prior cytotoxic therapies and the frequency of patients who survive progression-free for at least 6 months after initiating therapy or have objective tumor response.

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of adverse events as assessed by Common Terminology Criteria for Adverse Events version 4 (CTCAE v4) among women with leiomyosarcoma treated with MLN8237.

II. To determine the distribution of progression-free survival (PFS) and overall survival (OS).

TERTIARY OBJECTIVES:

I. To determine the relationship of Aurora A Kinase expression, measured by immunohistochemistry, with objective response, PFS at 6 months, survival, and progression-free survival.

OUTLINE:

Patients receive alisertib orally (PO) twice daily (BID) on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have incurable recurrent or persistent uterine leiomyosarcoma; histologic confirmation of the original primary tumor is required
* Patients must have measurable disease; measurable disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1); measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST version 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III protocol for the same patient population (12/10/2012)
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2; patients who have received two prior regimens must have a GOG performance status of 0 or 1
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
* Any other prior therapy directed at the malignant tumor, including chemotherapy and immunologic agents, must be discontinued at least three weeks prior to registration (12/10/2012)
* Any prior radiation therapy must be discontinued at least four weeks prior to registration (12/10/2012)
* Patients must have had at least one prior chemotherapeutic regimen for management of leiomyosarcoma
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease (12/10/2012)
* Patients must NOT have received any prior therapy directed at Aurora kinase for management of recurrent or persistent disease; patients who were treated on GOG-0250 (gemcitabine + docetaxel plus bevacizumab vs placebo) are eligible; treatment on GOG-0250 would count as ONE prior regimen
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Serum creatinine =< institutional upper limit of normal (ULN) OR creatinine clearance >= 60 mL/min/1.73m^2 (calculated or measured)
* Bilirubin =< ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception; pregnant women are excluded from this study
* Patients must be able to take oral medication and to maintain a fast for 2 hours before and 1 hour after MLN8237 administration
* Patient must not have taken agents that effect gastric pH within 4 days (any proton pump inhibitor), or 1 day (any histamine-2 antagonist) of the planned start of therapy; patients must be able to avoid all other types of antacids for 2 hours before and 2 hours after each dose of MLN8237

Exclusion Criteria:

* Patients who have had prior therapy with MLN8237 or taken part in a study of an investigational compound or device within 4 weeks of entering this study
* Patients who have had surgery (excluding biopsy), radiotherapy, or chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to the planned start of protocol treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients who have had hormonal agents within 1 week of the planned start of protocol treatment
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, carcinoma in situ of the cervix, or ductal carcinoma in situ of the breast, are excluded if there is any evidence of other malignancy being present within the last three years
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of uterine leiomyosarcoma within the last three years are excluded; thus, patients with a history of prior pelvic radiation for uterine leiomyosarcoma are eligible; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of uterine leiomyosarcoma within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients who are nursing because there is an unknown but potential risk for adverse events in nursing infants from MLN8237
* Patients with a history of central nervous system metastases and/or carcinomatous meningitis
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN8237, including but not limited to established allergic reaction to benzodiazepines
* Patients who are known to be human immunodeficiency virus (HIV) positive
* Patients who have had prior allogeneic bone marrow or organ transplantation
* Patients with a known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen; or any conditions that could result in excessive toxicity associated with the benzodiazepine-like effects of MLN8237
* Patients who require constant administration of proton pump inhibitor, H2 antagonist, or pancreatic enzymes; intermittent uses of antacids or H2 antagonists are allowed
* Patients who are unable to swallow oral medication or to maintain a fast as required for 2 hours before and 1 hour after MLN8237 administration or any condition that would modify small bowel absorption of oral medications, including malabsorption, or resection of pancreas or upper bowel
* Patients who have had treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine, oxcarbazepine, primidone or phenobarbital, or rifampin, rifabutin, rifapentine, or St. John's wort within 14 days prior to the first dose of MLN8237 and during the study
* Patients who have had a myocardial infarction within 6 months prior to enrollment or have New York Heart Association (NYHA) class III (marked limitation of physical activity, comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea) or IV (unable to carry out any physical activity without discomfort, symptoms of cardiac insufficiency at rest, if any physical activity is undertaken, discomfort is increased) heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Patients must limit alcohol consumption to no more than 1 standard unit of alcohol (12 oz beer [350 mL], 1.5 oz [45 mL] of 80-proof alcohol, or one 6-oz [175 mL] glass of wine) per day during the study and for 30 days from the last dose of MLN8237; patients who are unable to comply with these restrictions are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2017-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hyman, Principal Investigator — NRG Oncology
Locations (50):
- United States (50):
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Florida Hospital Orlando, Orlando, Florida
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Memorial Hermann Texas Medical Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 8/6/2012 and closed to accrual on 6/3/2013.
Groups:
- MLN8237: MLN8237, 50 mg, taken by mouth twice daily on Days 1-7. One cycle is 3 weeks long (21 days). CT or MRI imaging for response every other cycle (every 6 weeks). Treatment may continue until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | MLN8237
Started | 23
Completed | 21 (Eligible and treated patients.)
Not Completed | 2
Not completed — Ineligible: wrong primary | 1
Not completed — Ineligible: inadequate pathology | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | MLN8237
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.0)
Age, Customized [Number; unit: participants]
  40-49 years | 3
  50-59 years | 6
  60-69 years | 9
  70-79 years | 2
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
FIGO (International Federation of Gynecology and Obstetrics) Stage - Recurrent/Persistent [Number; unit: participants] | 21
Histologic Type - Leiomyosarcoma [Number; unit: participants] | 21

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) > 6 Months
Description: Whether or not the patient survived progression-free for at least 6 months. 90% confidence interval (Bonferroni Corrected). Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). Progression includes the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Assessed every other cycle for the first 6 months; then every 3 months from the date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | MLN8237
Number analyzed (Participants) | 21
percentage of participants | 0.0 [0.0 to 16.1]

2. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by RECIST 1.1. Patient response uses best overall response while on therapy. Complete response is defined as the disappearance of all target lesions and non-target lesions, and any pathological lymph nodes (whether target or non-target) must have reduction in the short axis to <10 mm. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete or partial response requires confirmation at greater than or equal to 4 weeks from initial documentation.
Time Frame: Every other cycle for the first 6 months; then every 3 months thereafter until withdrawal from study treatment or disease progression is confirmed.
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | MLN8237
Number analyzed (Participants) | 21
percentage of participants | 0.0 [0.0 to 16.1]

3. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years.
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MLN8237
Number analyzed (Participants) | 21
months | 13.6 [5.65 to 17.28]

4. Secondary Outcome: Number of Participants With Adverse Events as Assessed by NCI CTCAE Version 4.0
Time Frame: Every cycle during treatment and 30 days after the last treatment, up to 5 years.
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 4.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 4.0
- Grade 2 (CTCAE v 4.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 4.0
- Grade 3 (CTCAE v 4.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 4.0
- Grade 4 (CTCAE v 4.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 4.0
- Grade 5 (CTCAE v 4.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 4.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 4.0) | Grade 2 (CTCAE v 4.0) | Grade 3 (CTCAE v 4.0) | Grade 4 (CTCAE v 4.0) | Grade 5 (CTCAE v 4.0)
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 21 | 21
Participants
  Leukopenia | 9 | 3 | 4 | 5 | 0 | 0
  Thrombocytopenia | 11 | 9 | 0 | 1 | 0 | 0
  Neutropenia | 11 | 0 | 3 | 5 | 2 | 0
  Anemia | 5 | 3 | 9 | 3 | 1 | 0
  Other investigations | 18 | 3 | 0 | 0 | 0 | 0
  Other blood/lymphatics | 19 | 0 | 0 | 1 | 1 | 0
  Cardiac | 20 | 0 | 0 | 1 | 0 | 0
  Nausea | 15 | 3 | 3 | 0 | 0 | 0
  Vomiting | 18 | 3 | 0 | 0 | 0 | 0
  Other gastrointestinal | 4 | 7 | 6 | 4 | 0 | 0
  General and administration site | 9 | 5 | 7 | 0 | 0 | 0
  Infections/infestations | 19 | 0 | 2 | 0 | 0 | 0
  Metabolism/nutrition | 14 | 1 | 6 | 0 | 0 | 0
  Musculoskeletal/connective tissue | 16 | 3 | 1 | 1 | 0 | 0
  Peripheral sensory neuropathy | 20 | 1 | 0 | 0 | 0 | 0
  Nervous system | 12 | 5 | 4 | 0 | 0 | 0
  Psychiatric | 19 | 2 | 0 | 0 | 0 | 0
  Renal/urinary | 19 | 2 | 0 | 0 | 0 | 0
  Reproductive/breast | 19 | 1 | 0 | 1 | 0 | 0
  Respiratory/thoracic/mediastinal | 16 | 4 | 0 | 1 | 0 | 0
  Skin/subcutaneous | 7 | 5 | 7 | 2 | 0 | 0
  Vascular disorders | 19 | 0 | 1 | 1 | 0 | 0

5. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression was based on RECIST 1.1. RECIST 1.1 defines progressive disease as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions or unequivocal progression of non-target lesions is also considered progression.
Time Frame: every other cycle for the first 6 months; then every 3 months thereafter until disease progression is confirmed; up to 5 years
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | MLN8237
Number analyzed (Participants) | 21
months | 1.7 [1.4 to 3.2]

6. Other Pre Specified Outcome: Aurora A Kinase Expression
Description: Aurora A Kinase expression will be assessed for associations with patient demographics and clinical outcome (response, PFS at 6 months, PFS, and OS).
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) during treatment (up to 30 days after treatment completion). All Serious Adverse Events (SAEs) up to 30 days after treatment completion and considered to be treatment related between 30 days and 5 years after treatment completion.
Arm/Group | MLN8237
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN8237 (N=21)
Anemia (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN8237 (N=21)
Anemia (Blood and lymphatic system disorders) | 15
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 3
Stomach Pain (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Mucositis Oral (Gastrointestinal disorders) | 9
Oral Hemorrhage (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3
Esophagitis (Gastrointestinal disorders) | 1
Pain (General disorders) | 5
Localized Edema (General disorders) | 1
Fatigue (General disorders) | 13
Fever (General disorders) | 2
Chills (General disorders) | 1
Mucosal Infection (Infections and infestations) | 2
Vaginal Infection (Infections and infestations) | 1
Weight Loss (Investigations) | 1
Platelet Count Decreased (Investigations) | 10
Neutrophil Count Decreased (Investigations) | 10
White Blood Cell Decreased (Investigations) | 12
Aspartate Aminotransferase Increased (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Somnolence (Nervous system disorders) | 5
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hot Flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less